CLINICAL TRIAL: NCT06173947
Title: Spleen Stiffness Measurement Predicts Short-term Outcomes of Chronic Liver Disease Inpatients With Acute Liver Injury: a Prospective, Observational and Multicentre Study
Brief Title: SSM Predicts Outcomes of CLD Inpatients With Acute Liver Injury
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-495
Record Dates: First submitted 2023-11-24; First posted 2023-12-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: End Stage Liver Disease; Jaundice; Liver Dysfunction; Portal Hypertension
Keywords: End Stage Liver Disease; Chronic Liver Disease; Spleen Stiffness Measurement; Acute-on-Chronic Liver Failure; Portal Hypertension; Jaundice
MeSH Terms: conditions — End Stage Liver Disease; Jaundice; Liver Diseases; Hypertension, Portal; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will collect biospecimens, including whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FibroScan® Expert 630 — The SSM by FibroScan 630 was first performed after admission, repeated at the day 5±2 as soon as feasible, and finally evaluated before discharge.
  Other Names: FibroScan® (FibroScan® expert 630 machine; Echosens, Paris, France); Spleen mode (SSM@100 Hz); Spleen vibration-controlled transient elastography (VCTE) settings (SSM@100 Hz); Spleen-dedicated examination based on VCTE (SSM@100 Hz)

SUMMARY:
In this study, a single non-invasive tool, spleen stiffness measurement (SSM), was used to monitor the disease regression of inpatients with chronic liver disease (CLD) and acute liver injury. The present study aimed to establish an early diagnosis warning model for acute-on-chronic liver failure (ACLF) by SSM and investigate the effect of dynamic changes in SSM on the short-term prognosis (28-day, 90-day morbidity and mortality) of inpatients with CLD and acute liver injury.

DETAILED DESCRIPTION:
Portal hypertension is a major complication of cirrhosis and can lead to serious clinical manifestations such as ascites, hepatic encephalopathy, variceal bleeding, etc. Colecchia et al. proposed the use of spleen stiffness measurement (SSM) to dynamically monitor portal pressure and to predict the risk of oesophageal varices. Studies have now demonstrated the utility of SSM in assessing portal hypertension, ruling out high-risk varices, and predicting clinical complications in cirrhotic patients. Furthermore, the Baveno VII consensus of portal hypertension has included SSM in its recommendations for non-invasive screening. Pathogenic triggers, important clinical events (ascites, encephalopathy, etc.), and short-term prognosis in compensated advanced chronic liver disease are associated with portal pressure. Exploring the relationship between portal hypertension and liver failure development would be of great clinical and scientific value. The present study is mainly based on a single non-invasive tool, SSM, to monitor the disease regression of chronic liver disease (CLD) inpatients with acute liver injury, to establish an early warning model for early diagnosis of acute-on-chronic liver failure, and to investigate the effect of dynamic changes in SSM on the short-term prognosis of inpatients with CLD and acute liver injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years and 80 years
2. Chronic liver diseases regardless of etiology
3. Acute liver injury with total bilirubin ≥ 3 mg/dl regardless of inducement

Exclusion Criteria:

1. Prior surgery of liver diseases before enrollment such as liver transplantation, transjugular intrahepatic portosystemic shunt (TIPS), splenectomy and partial splenic embolization
2. Severe extrahepatic diseases such as chronic obstructive pulmonary disease level IV, chronic kidney disease with end-stage renal failure, myocardial infarction within 3 months before admission
3. Receiving Immunosuppressive drugs for reasons rather than chronic liver diseases
4. Diagnosis of hepatocellular carcinoma or other non-liver malignancies during screening period
5. Serious mental illnesses such as anxiety, depressive disorders to obsessive-compulsive disorder (OCD) and post-traumatic stress disorder (PTSD)
6. The pregnant
7. Jaundice due to biliary obstruction or cholestasis
8. Unsuitable to participate in this study judging by investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cirrhosis or other chronic liver diseases and hospitalized for acute liver injury with total bilirubin [TB] ≥3 mg/dl were admitted.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
90-day transplant-free mortality | Day 90
  The primary endpoint was 90-day transplant-free mortality, defined as all-cause death within 90 days, including deaths within the initial hospitalization, after discharge, after transfer to other acute care facilities, and requiring readmission.

SECONDARY OUTCOMES:
Incidence of acute kidney injury (AKI) | From admission to Day 90
  AKI is defined as a change in SCr of ≥ 0.3 mg/dl (26.5 μmol/L) in ≤ 48 h, or a 50% increase in SCr from a baseline that is known or presumed to have occurred in the past 7 days.
Rate of progression to acute-on-chronic liver failure (ACLF) | From admission to Day 90
  ACLF was defined according to the European Association for the Study of Liver-Chronic Liver Failure (EASL-CLIF) criteria. ACLF grade-1 includes three subgroups: 1) patients with single kidney failure; 2) patients with single failure of the liver, coagulation, circulation or respiration, who had serum creatinine ranging from 1.5 to 1.9 mg/dl and/or mild-to-moderate hepatic encephalopathy; and 3) patients with single cerebral failure who had serum creatinine ranging from 1.5 and 1.9 mg/dl. ACLF grade-2: patients with two organs failure. ACLF grade-3: patients with three organ failures or more. ACLF development: patients with absence of ACLF on admission and progression to ACLF within 28 days. The severity of liver disease was evaluated by the model of end-stage liver disease (MELD) score, Child-Pugh score and CLIF-AD score (in those without ACLF).
Rate for readmission of patients hospitalized with acute liver injury | From discharge to Day 90
  The readmission was rehospitalization with liver-related complications (including bacterial infection, variceal bleeding, overt hepatic encephalopathy, or a new onset or worsening of ascites) at any ward to any hospital in the following discharge from the index admission with acute liver injury.

CONTACTS AND LOCATIONS:
Overall Officials: Jinjun Chen, PHD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Use a public management platform for clinical trials and make it accessible to the public, or contact the investigator for primary data by E-mail.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The deidentified individual patient data (IPD) underlying the results presented in the article (including tables, figures, and appendices or supplementary material) no later than six months after publication.
Access Criteria: Data will be made available on request from the corresponding author.

REFERENCES:
- [Result] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Result] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Result] Moreau R, Jalan R, Gines P, Pavesi M, Angeli P, Cordoba J, Durand F, Gustot T, Saliba F, Domenicali M, Gerbes A, Wendon J, Alessandria C, Laleman W, Zeuzem S, Trebicka J, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Acute-on-chronic liver failure is a distinct syndrome that develops in patients with acute decompensation of cirrhosis. Gastroenterology. 2013 Jun;144(7):1426-37, 1437.e1-9. doi: 10.1053/j.gastro.2013.02.042. Epub 2013 Mar 6. PMID 23474284
- [Result] Wu T, Li J, Shao L, Xin J, Jiang L, Zhou Q, Shi D, Jiang J, Sun S, Jin L, Ye P, Yang L, Lu Y, Li T, Huang J, Xu X, Chen J, Hao S, Chen Y, Xin S, Gao Z, Duan Z, Han T, Wang Y, Gan J, Feng T, Pan C, Chen Y, Li H, Huang Y, Xie Q, Lin S, Li L, Li J; Chinese Group on the Study of Severe Hepatitis B (COSSH).. Development of diagnostic criteria and a prognostic score for hepatitis B virus-related acute-on-chronic liver failure. Gut. 2018 Dec;67(12):2181-2191. doi: 10.1136/gutjnl-2017-314641. Epub 2017 Sep 19. PMID 28928275
- [Result] Li J, Liang X, You S, Feng T, Zhou X, Zhu B, Luo J, Xin J, Jiang J, Shi D, Lu Y, Ren K, Wu T, Yang L, Li J, Li T, Cai Q, Sun S, Guo B, Zhou X, Chen J, He L, Li P, Yang H, Hu W, An Z, Jin X, Tian J, Wang B, Chen X, Xin S, Li J; Chinese Group on the Study of Severe Hepatitis B (COSSH). Development and validation of a new prognostic score for hepatitis B virus-related acute-on-chronic liver failure. J Hepatol. 2021 Nov;75(5):1104-1115. doi: 10.1016/j.jhep.2021.05.026. Epub 2021 Jun 4. PMID 34090929
- [Result] de Franchis R, Pascal JP, Ancona E, Burroughs AK, Henderson M, Fleig W, Groszmann R, Bosch J, Sauerbruch T, Soederlund C, et al. Definitions, methodology and therapeutic strategies in portal hypertension. A Consensus Development Workshop, Baveno, Lake Maggiore, Italy, April 5 and 6, 1990. J Hepatol. 1992 May;15(1-2):256-61. doi: 10.1016/0168-8278(92)90044-p. No abstract available. PMID 1506645
- [Result] Karagiannakis DS, Voulgaris T, Siakavellas SI, Papatheodoridis GV, Vlachogiannakos J. Evaluation of portal hypertension in the cirrhotic patient: hepatic vein pressure gradient and beyond. Scand J Gastroenterol. 2018 Oct-Nov;53(10-11):1153-1164. doi: 10.1080/00365521.2018.1506046. Epub 2018 Oct 21. PMID 30345856
- [Result] Berzigotti A, Bosch J, Boyer TD. Use of noninvasive markers of portal hypertension and timing of screening endoscopy for gastroesophageal varices in patients with chronic liver disease. Hepatology. 2014 Feb;59(2):729-31. doi: 10.1002/hep.26652. Epub 2013 Dec 24. No abstract available. PMID 23913844
- [Result] Vizzutti F, Arena U, Romanelli RG, Rega L, Foschi M, Colagrande S, Petrarca A, Moscarella S, Belli G, Zignego AL, Marra F, Laffi G, Pinzani M. Liver stiffness measurement predicts severe portal hypertension in patients with HCV-related cirrhosis. Hepatology. 2007 May;45(5):1290-7. doi: 10.1002/hep.21665. PMID 17464971
- [Result] Colecchia A, Montrone L, Scaioli E, Bacchi-Reggiani ML, Colli A, Casazza G, Schiumerini R, Turco L, Di Biase AR, Mazzella G, Marzi L, Arena U, Pinzani M, Festi D. Measurement of spleen stiffness to evaluate portal hypertension and the presence of esophageal varices in patients with HCV-related cirrhosis. Gastroenterology. 2012 Sep;143(3):646-654. doi: 10.1053/j.gastro.2012.05.035. Epub 2012 May 27. PMID 22643348
- [Result] Colecchia A, Colli A, Casazza G, Mandolesi D, Schiumerini R, Reggiani LB, Marasco G, Taddia M, Lisotti A, Mazzella G, Di Biase AR, Golfieri R, Pinzani M, Festi D. Spleen stiffness measurement can predict clinical complications in compensated HCV-related cirrhosis: a prospective study. J Hepatol. 2014 Jun;60(6):1158-64. doi: 10.1016/j.jhep.2014.02.024. Epub 2014 Mar 6. PMID 24607624
- [Result] Berzigotti A. Non-invasive evaluation of portal hypertension using ultrasound elastography. J Hepatol. 2017 Aug;67(2):399-411. doi: 10.1016/j.jhep.2017.02.003. Epub 2017 Feb 14. PMID 28223101
- [Result] Colecchia A, Ravaioli F, Marasco G, Colli A, Dajti E, Di Biase AR, Bacchi Reggiani ML, Berzigotti A, Pinzani M, Festi D. A combined model based on spleen stiffness measurement and Baveno VI criteria to rule out high-risk varices in advanced chronic liver disease. J Hepatol. 2018 Aug;69(2):308-317. doi: 10.1016/j.jhep.2018.04.023. Epub 2018 May 3. PMID 29729368
- [Result] Wang H, Wen B, Chang X, Wu Q, Wen W, Zhou F, Guo Y, Ji Y, Gu Y, Lai Q, He Q, Li J, Chen J, Hou J. Baveno VI criteria and spleen stiffness measurement rule out high-risk varices in virally suppressed HBV-related cirrhosis. J Hepatol. 2021 Mar;74(3):584-592. doi: 10.1016/j.jhep.2020.09.034. Epub 2020 Oct 8. PMID 33039403
- [Result] Stefanescu H, Marasco G, Cales P, Fraquelli M, Rosselli M, Ganne-Carrie N, de Ledinghen V, Ravaioli F, Colecchia A, Rusu C, Andreone P, Mazzella G, Festi D. A novel spleen-dedicated stiffness measurement by FibroScan(R) improves the screening of high-risk oesophageal varices. Liver Int. 2020 Jan;40(1):175-185. doi: 10.1111/liv.14228. Epub 2019 Sep 11. PMID 31444849
- [Result] Reiberger T. The Value of Liver and Spleen Stiffness for Evaluation of Portal Hypertension in Compensated Cirrhosis. Hepatol Commun. 2022 May;6(5):950-964. doi: 10.1002/hep4.1855. Epub 2021 Dec 14. PMID 34904404
- [Result] Zhang X, Song J, Zhang Y, Wen B, Dai L, Xi R, Wu Q, Li Y, Luo X, Lan X, He Q, Luo W, Lai Q, Ji Y, Zhou L, Qi T, Liu M, Zhou F, Wen W, Li H, Liu Z, Chen Y, Zhu Y, Li J, Huang J, Cheng X, Tu M, Hou J, Wang H, Chen J. Baveno VII algorithm outperformed other models in ruling out high-risk varices in individuals with HBV-related cirrhosis. J Hepatol. 2023 Mar;78(3):574-583. doi: 10.1016/j.jhep.2022.10.030. Epub 2022 Nov 7. PMID 36356684
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines for the management of patients with decompensated cirrhosis. J Hepatol. 2018 Aug;69(2):406-460. doi: 10.1016/j.jhep.2018.03.024. Epub 2018 Apr 10. No abstract available. PMID 29653741
- [Result] Sarin SK, Choudhury A, Sharma MK, Maiwall R, Al Mahtab M, Rahman S, Saigal S, Saraf N, Soin AS, Devarbhavi H, Kim DJ, Dhiman RK, Duseja A, Taneja S, Eapen CE, Goel A, Ning Q, Chen T, Ma K, Duan Z, Yu C, Treeprasertsuk S, Hamid SS, Butt AS, Jafri W, Shukla A, Saraswat V, Tan SS, Sood A, Midha V, Goyal O, Ghazinyan H, Arora A, Hu J, Sahu M, Rao PN, Lee GH, Lim SG, Lesmana LA, Lesmana CR, Shah S, Prasad VGM, Payawal DA, Abbas Z, Dokmeci AK, Sollano JD, Carpio G, Shresta A, Lau GK, Fazal Karim M, Shiha G, Gani R, Kalista KF, Yuen MF, Alam S, Khanna R, Sood V, Lal BB, Pamecha V, Jindal A, Rajan V, Arora V, Yokosuka O, Niriella MA, Li H, Qi X, Tanaka A, Mochida S, Chaudhuri DR, Gane E, Win KM, Chen WT, Rela M, Kapoor D, Rastogi A, Kale P, Rastogi A, Sharma CB, Bajpai M, Singh V, Premkumar M, Maharashi S, Olithselvan A, Philips CA, Srivastava A, Yachha SK, Wani ZA, Thapa BR, Saraya A, Shalimar, Kumar A, Wadhawan M, Gupta S, Madan K, Sakhuja P, Vij V, Sharma BC, Garg H, Garg V, Kalal C, Anand L, Vyas T, Mathur RP, Kumar G, Jain P, Pasupuleti SSR, Chawla YK, Chowdhury A, Alam S, Song DS, Yang JM, Yoon EL; APASL ACLF Research Consortium (AARC) for APASL ACLF working Party.. Acute-on-chronic liver failure: consensus recommendations of the Asian Pacific association for the study of the liver (APASL): an update. Hepatol Int. 2019 Jul;13(4):353-390. doi: 10.1007/s12072-019-09946-3. Epub 2019 Jun 6. PMID 31172417